CLINICAL TRIAL: NCT00140166
Title: The Treatment of Acute Schizophrenia With High Dose Niacinmide Plus Ascorbate Plus Pyridoxine Plus Centrum Forte vs. Centrum Forte Only as an Add-On to Risperidone and Dietary Counseling
Brief Title: Treatment of Acute Schizophrenia With Vitamin Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beersheva Mental Health Center (Other Government)
Collaborators: Supported by a Hilton Family Foundation grant to (Unknown); International Schizophrenia Foundation (Unknown)
Responsible Party: Vladimir Lerner, Ben Gurion University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMHC-3996
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Acute Schizophrenia
Keywords: schizophrenia; niacinamide
MeSH Terms: conditions — Schizophrenia | interventions — Niacinamide; Pyridoxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: niacinamide
Drug: pyridoxine
Drug: ascorbate

SUMMARY:
Controlled studies using the orthomolecular approach have been few (Deutsch, Ananth, & Ban, 1977). Those that were done were performed in chronic schizophrenia or in populations that included bipolar and schizoaffective patients. Both of these diagnostic groups are not today considered to benefit from the orthomolecular approach. Moreover, some negative studies of high-dose niacin were done in patients who were not otherwise given general counseling for good diet as described above. Therefore, this proposal is to study in a controlled manner carefully defined first onset schizophrenic patients using the protocol advocated by Osmond and Hoffer (1962). Patients can enter the study if they have been ill less than 1 year and are in their first hospitalization.

DETAILED DESCRIPTION:
Controlled studies using the orthomolecular approach have been few (Deutsch, Ananth, & Ban, 1977). Those that were done were performed in chronic schizophrenia or in populations that included bipolar and schizoaffective patients. Both of these diagnostic groups are not today considered to benefit from the orthomolecular approach. Moreover, some negative studies of high-dose niacin were done in patients who were not otherwise given general counseling for good diet as described above. Therefore, this proposal is to study in a controlled manner carefully defined first onset schizophrenic patients using the protocol advocated by Osmond and Hoffer (1962). Patients can enter the study if they have been ill less than 1 year and are in their first hospitalization. Our Beersheba Mental Health Center is the only hospitalization facility for Southern Israel, population of half a million. There about 2 thousand admissions to our hospital yearly and of those there are over 100 admissions with a diagnosis of schizophrenia or schizophreniform disorder for whom this is the first lifetime admission to hospital and their first episode of psychosis.

Methods Study I - Open Pilot The pilot study will be carried out exactly as below, except without a control group. Results from the pilot will be evaluated before continuing to the controlled study, and protocol modifications presented to the Helsinki Committee if necessary. Ten patients will be studied in this open pilot study.

Study II - Controlled Study, Not Blind Inclusion and exclusion criteria Patients can be accepted to the study age 18-30, if admitting diagnosis after review by the study coordinator is schizophrenia or schizophreniform disorder by DSM-IV. Since the diagnosis of schizophrenia may be difficult in the early stages of acute psychotic disease, cases in which the clinical diagnosis is consistent with and suspicious of schizophrenia (and inconsistent with bipolar disorder) even if they do not fulfill all the diagnostic criteria in DSM-IV will be accepted. Patients with alcohol or drug abuse in the last 6 months will be excluded. Patients with significant physical illness including peptic ulcer, or a history of hepatitis or baseline abnormal liver function tests will be excluded. Patients with mental retardation will be excluded. Baseline screening will be done for liver function (including AST, bilirubin, alkaline phosphatase and LDH) and blood glucose and then repeated after 6 weeks. Elevations of AST over three fold will lead to dropping patient from study. Patients who are unlikely to be able to continue in the study as outpatients will be excluded. Patients will be admitted to study only if this is their first lifetime psychiatric admission and their first episode of psychosis and only if history supports that they have been mentally ill for less than one year.

Procedure Patients who enter the program will be treated with risperidone, 2-8mg daily at physician's discretion . They will be randomized according to a predetermined random order to vitamin regime or Centrum forte. Doses of risperidone will be lowered as clinically possible. Risperidone dose will be recorded weekly and will serve as a secondary outcome measure. A registered dietician will meet with each patient weekly and discourage refined sugar or excess fat and encourage regular fruit and vegetable consumption. High protein breakfast will be emphasized. Fifteen patients will be started yearly for three years.

The vitamin regimen will be as follows twice daily with food:

1. Ascorbic acid 1.5 g twice daily.
2. 150 mg vitamin B6 twice daily
3. Niacinamide 500 mg tablets, 3 tablets (1.5g) twice daily with food.
4. Centrum Forte, one tablet each morning with food.

The comparison group will receive Centrum Forte once per day.

Outcome measures

Patients will be rated with the Brief Psychiatric Rating Scale (BPRS) at baseline and weekly for 6 months. All patients will receive supportive psychotherapy both during the hospitalization and in clinic follow-up. Discharged patients will be followed in the outpatient clinic of the Beersheba Mental Health Center by a physician plus dietician team dedicated to this study. Each patient will be followed for six months. Outcome measures will be BPRS ratings over the course of the half year, readmissions, Global Clinical Assessment of function at the end of the half year, and risperidone dose.

Skin test A blunted response of dermal erythema to niacin has been widely reported in schizophrenia, and it is possible that this response might predict clinical response to niacin treatment. All patients will have the Horrobin niacin patch test (Smesny et al., 2003) on admission to the study and it will be repeated after 6 months of continuous therapy. Niacin is applied simultaneously in four dilutions (0.1, 0.01, 0.001, 0.0001M) of 50microl each (approximately one drop of a standard eye-dropper) to the skin at the inner side of the forearm using chambered plaster for epicutaneous testing. After 90 seconds the plaster is removed. Skin reaction is quantitated at 3 minute intervals up to 21 minutes starting 90 seconds after removal of the plaster.

Risks The risks of high dose ascorbic acid have been reviewed extensively but these refer to doses such as 10g daily and the present dose of 3g daily is associated with minimal risk eg diarrhea. Doses greater than 3gm daily can cause increases in ALT and uric acid but risk of kidney stones has not been substantiated (Russel, 2005). Niacin at 3g daily is now widely used as a cholesterol lowering agent (Alpers, Stenson, & Bier, 2002) and is associated with minimal side effects or dangers eg, up to 5% increased glucose, elevations of liver enzymes and exacerbation in peptic ulcer, but these effects are rarely if ever seen with the derivative nicotinamide (Guyton, 2005). The other B-vitamins in the doses given would not be associated with any side effects.

Alpers, D. H., Stenson, W. F., & Bier, D. M. (2002). Manual of Nutritional Therapeutics. Philadelphia: Lippincott Williams & Wilkins.

Beauclair, L., Vinogradov, S., Riney, S. J., Csernansky, J. G., & Hollister, L. E. (1987). An adjunctive role for ascorbic acid in the treatment of schizophrenia? J Clin Psychopharmacol, 7(4), 282-283.

Deutsch, M., Ananth, J. V., & Ban, T. A. (1977). Nicotinic acid in the treatment of chronic hospitalized schizophrenic patients: a placebo-controlled clinical study. Psychopharmacol Bull, 13(3), 21-23.

Guyton, J. R. (2005). Hyperlimpprotenemias. In R. E. Rakel & E. T. Bope (Eds.), Conn's Current Therapy 2005 (pp. 688-694). Pennsylvania: Elsevier/Saunders.

Kanofsky, J. D., & Sandyk, R. (1992). Antioxidants in the treatment of schizophrenia. Int J Neurosci, 62(1-2), 97-100.

Kleijnen, J., & Knipschild, P. (1991). Niacin and vitamin B6 in mental functioning: a review of controlled trials in humans. Biol Psychiatry, 29(9), 931-941.

Lerner, V., Miodownik, C., Kaptsan, A., Cohen, H., Loewenthal, U., & Kotler, M. (2002). Vitamin B6 as add-on treatment in chronic schizophrenic and schizoaffective patients: a double-blind, placebo-controlled study. J Clin Psychiatry, 63(1), 54-58.

Levine, J., Stahl, Z., Sela, B. A., Ruderman, V., Shumaico, O., Babushkin, I., et al. (under revision). Homocysteine reducing strategies improve symptoms in chronic schizophrenia patients with hyperhomocysteinemia.

Osmond, H., & Hoffer, A. (1962). Massive niacin treatment in schizophrenia. Review of a nine-year study. Lancet, 1, 316-319.

Russel, R. M. (2005). Vitamine and trace mineral deficiency and excess. In D. L. Kasper, A. S. Favci, D. L. Lango, E. Braunwald, S. L. Hauser & J. L. Jameson (Eds.), Harrison's Principles of Internal Medicine (16th ed., pp. 403-407): McGraw Hill.

Sandyk, R., & Kanofsky, J. D. (1993). Vitamin C in the treatment of schizophrenia. Int J Neurosci, 68(1-2), 67-71.

Smesny, S., Berger, G., Rosburg, T., Riemann, S., Riehemann, S., McGorry, P., et al. (2003). Potential use of the topical niacin skin test in early psychosis -- a combined approach using optical reflection spectroscopy and a descriptive rating scale. J Psychiatr Res, 37(3), 237-247.

Smythies, J. R. (1996). The role of ascorbate in brain: therapeutic implications. J R Soc Med, 89(5), 241..

Straw, G. M., Bigelow, L. B., & Kirch, D. G. (1989). Haloperidol and reduced haloperidol concentrations and psychiatric ratings in schizophrenic patients treated with ascorbic acid. J Clin Psychopharmacol, 9(2), 130-132.

Suboticanec, K., Folnegovic-Smalc, V., Korbar, M., Mestrovic, B., & Buzina, R. (1990). Vitamin C status in chronic schizophrenia. Biol Psychiatry, 28(11), 959-966.

Suboticanec, K., Folnegovic-Smalc, V., Turcin, R., Mestrovic, B., & Buzina, R. (1986). Plasma levels and urinary vitamin C excretion in schizophrenic patients. Hum Nutr Clin Nutr, 40(6), 421-428.

Vaughan, K., & McConaghy, N. (1999). Megavitamin and dietary treatment in schizophrenia: a randomised, controlled trial. Aust N Z J Psychiatry, 33(1), 84-88.

ELIGIBILITY:
Inclusion Criteria:

* age 18-30
* schizophrenia or schizophreniform disorder
* first psychiatric admission and first episode of psychosis
* mentally ill for less than one year

Exclusion Criteria:

* alcohol or drug abuse in last 6 months
* significant physical illness
* mental retardation

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2005-07; Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Brief Psychiatric Rating Scale
Global Clinical Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Lerner, MD, Principal Investigator — Beersheva Mental Health Center; RH Belmaker, MD, Study Director — Ben-Gurion University of the Negev
Locations (1):
- Beersheva Mental Health Center, Beersheva, Israel